CLINICAL TRIAL: NCT05595109
Title: The Possible Protective Role of Silymarin Against Chemotherapy Induced Toxicities and Cognitive Impairment in Breast Cancer Patients
Brief Title: Role of Silymarin in Chemotherapy Toxicity and Cognition Improvement in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Azza Ahmed Abdelkader Abu El-atta, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35945/10/22
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Peripheral Neuropathy; Cardiac Toxicities; Hepatic Toxicity; Cognitive Impairment
Keywords: Breast Cancer; neuropathy; Cardiac Toxicities; Hepatic Toxicity; Cognitive Impairment; Chemotherapy; Toxicities; Silymarin
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases; Cardiotoxicity; Cognitive Dysfunction | interventions — Silymarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group one: (Placebo group) (Placebo Comparator): which will receive four cycles of AC regimen (doxorubicin and cyclophosphamide; each cycle was given every 21 day)
  followed by 12 cycles of paclitaxel (each cycle was given in a weekly basis) plus placebo tablets once daily.
  Interventions: Drug: Placebo
- Group two: (Silymarin group) (Active Comparator): which will receive the same regimen plus silymarin 140mg once daily.
  Interventions: Drug: Silymarin

INTERVENTIONS:
Drug: Silymarin — Silymarin administration prevent the neuro-degeneration through inhibiting the activation of microglia, silymarin attenuates the activation of glial cell activation in cellular models possibly through inhibition of inducible nitric oxide synthase (iNOS) production, also reported to protect both microglia and astroglia from oxidative insults induced by peroxide in ex vivo system .
  It also significantly reduces doxorubicin-pro-oxidative activity and decreases histological changes in liver and heart tissue . The hepato-protective and cardio-protective effects of silymarin may be attributed to its antioxidant capacity, its ability to prevent lipid peroxidation and its ability to increase glutathione concentration.
  silymarin was reported to improve cognitive impairment in mice.
  Arms: Group two: (Silymarin group)
Drug: Placebo — which will receive four cycles of AC regimen (doxorubicin and cyclophosphamide; each cycle was given every 21 day) followed by 12 cycles of paclitaxel (each cycle was given in a weekly basis) plus placebo tablets once daily.
  Arms: Group one: (Placebo group)

SUMMARY:
Aim of the work This study aims to evaluate the possible beneficial role of silymarin in attenuating both doxorubicin related cardiac and hepatic toxicities and paclitaxel associated peripheral neuropathy and improving cognitive impairment in patients with breast cancer.

This study will be a randomized placebo controlled parallel study. The study will be performed in accordance with the ethical standards of Helsinki declaration in 1964 and its later amendments.

Group one: (Placebo group; n=28) which will receive four cycles of AC regimen (doxorubicin and cyclophosphamide; each cycle was given every 21 day) followed by 12 cycles of paclitaxel (each cycle was given in a weekly basis) plus placebo tablets once daily.

Group two: (Silymarin group; n=28) which will receive the same regimen plus silymarin 140mg once daily

DETAILED DESCRIPTION:
Breast cancer represents the most frequently diagnosed malignancy and the second most common cause of cancer death worldwide. In Egypt, breast cancer is the most common malignancy in women, accounting for 38.8% of cancers in this population, with the estimated number of breast cancer cases nearly 22,700 in 2020 and forecasted to be approximately 46,000 in 2050 .

Paclitaxel and doxorubicin are cytotoxic agents that are commonly used for treatment of breast cancer. Despite their effectiveness, both paclitaxel and doxorubicin are associated with cumulative and potential neurotoxicity and cardiotoxicity respectively . Paclitaxel induced peripheral neuropathy (PN) is a consequence of activation of the inflammatory cascade with subsequent increased pro-inflammatory cytokines production including tumor necrosis factor-α (TNF-α), interleukin-1β (IL-1β) and interleukin-6 (IL-6) . Moreover, paclitaxel can up-regulate matrix metalloproteinase-3 (MMP3) which plays an important role in the inflammatory and degenerative processes following nerve injury .

Oxidative stress plays a critical role in doxorubicin associated cardiotoxicity through direct cellular damage, induction of apoptosis and activation of nuclear factor- Kabba B (NF-ĸB) which in turn stimulates the production and release of inflammatory mediators .

Hepatotoxicity from doxorubicin was reported and it is likely due to direct toxic injury to the liver. Doxorubicin and its analogues are metabolized in the liver via microsomal enzymes, and production of a toxic or immunogenic intermediate may trigger liver injury with subsequent elevation of Serum aminotransferase.In addition, it was reported that, doxorubicin related hepatotoxicity is a consequence of free radical formation and oxidative stress and antioxidants may protect against doxorubicin-induced toxicity in the liver .

Although, the underlying neuro-protective mechanism of silymarin is mainly due to its capacity to inhibit oxidative stress in the brain, it also confers additional neuro-protection by influencing other pathways such as inflammatory pathways . Silymarin has been implicated in protecting neurons against oxidative stress and nitrosative stress . Silymarin was reported to exert direct effect on neuronal oxidant status .

Silymarin administration in a lipopolysaccharide induced animal model of peripheral neuropathy prevented the dopaminergic neuro-degeneration through inhibiting the activation of microglia. Other in-vitro studies revealed that, silymarin attenuates the activation of glial cell activation in cellular models possibly through inhibition of inducible nitric oxide synthase (iNOS) production . Silymarin was also reported to protect both microglia and astroglia from oxidative insults induced by peroxide in ex vivo system .

Treatment with silymarin prevents the increase in AST and creatine kinase (CK) serum activity and myocardial excitability in rats caused by doxorubicin . It also significantly reduces doxorubicin-pro-oxidative activity and decreases histological changes in liver and heart tissue . The hepato-protective and cardio-protective effects of silymarin may be attributed to its antioxidant capacity, its ability to prevent lipid peroxidation and its ability to increase glutathione concentration .

Cognitive impairment in patients with breast cancer began to appear in the literature in the 1990s, coincident with the increasing use of postoperative adjuvant chemotherapy . In two recent preclinical studies, silymarin was reported to improve cognitive impairment in mice, and these former studies suggested that silymarin may be a therapeutic agent for cognitive decline .

This study will be a randomized placebo controlled parallel study. The study will be performed in accordance with the ethical standards of Helsinki declaration in 1964 and its later amendments.

Group one: (Placebo group; n=28) which will receive four cycles of AC regimen (doxorubicin and cyclophosphamide; each cycle was given every 21 day) followed by 12 cycles of paclitaxel (each cycle was given in a weekly basis) plus placebo tablets once daily.

Group two: (Silymarin group; n=28) which will receive the same regimen plus silymarin 140mg once daily.

* Blood sample collection and biochemical assessment:

  1. N-terminal prohormone of brain naturetic peptide (NT-proBNP" ) and liver panel.
  2. myeloperoxidase (MPO)
  3. neurofilament light chain (NFL)
  4. andnuclear factor- Kabba B p65 (NF-ĸB p65) or TNF-alpha
* Clinical assessment of chemotherapy induced toxicities:
* Doxorubicin related cardiotoxicity will be assessed through - Echocardiography at baseline and after the last doxorubicin/ cyclophosphamide (AC) cycle.
* Paclitaxel induced peripheral sensory neuropathy will be done through: - The implication of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017) for grading of neuropathy at baseline and by the end of every two paclitaxel cycles.
* The use of Neurotoxicity- 12 item questionnaire score (Ntx-12) from the validated Functional Assessment of Cancer Therapy/Gynecologic Oncology Group "FACT/GOG-Ntx-12" at baseline and by the end of every two paclitaxel cycles.
* The assessment of the severity of neuropathic pain through brief pain inventory short form "BPI-SF" worst item. Severity of neuropathic pain will be assessed at baseline and by the end of every two paclitaxel cycles.
* Cognitive impairment will be assessed using the brief assessment of impaired Cogentin questionnaire (BASIC-Q).
* Primary and secondary outcomes:

The primary outcome is the change in ejection fraction and percentage of patients with peripheral sensory neuropathy grade ≥ 2 with the variation of both 12-item neurotoxicity questionnaire (Ntx-12) total score and pain rating scale score. The secondary outcome is the changes in serum levels of the measured biological markers.

- Sample size calculation: According to the results of a previous study, the total number of subjects required to detect the cardio-protective effect of silymarin in patients with different types of cancer receiving anthracyclines containing chemotherapy was 25 patients . With 5% significance level, 80% statistical power and an attrition rate of 10%, the initial sample size required for the current study is 28 patients in each group.

-Ethical approval: The study will be approved by the Research Ethics Committee of Tanta University. The study will be registered as a clinical trial at ClinicalTrials.gov. All participants will be informed about the benefits and risks of the study. Any unexpected risks that will appear during the course of the research will be clarified to the participants and to the ethical committee on time. The data of the enrolled patients will be confidential. All enrolled patients will give their written informed consents. The study will be conducted between October 2022 and October 2024.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Patients with biopsy confirmed diagnosis breast cancer and with stage II and stage III breast cancer according to the American Joint Committee on Cancer (TNM staging system of breast cancer).
* Patients with performance status <2 according to Eastern Cooperative Oncology Group (ECOG) score.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate liver function (serum bilirubin < 1.2 mg/dl) and adequate renal function (serum creatinine< 1.5 mg/d).

Exclusion Criteria:

* Patients with prior exposure to anthracyclines and neurotoxic agents (Cis-platin, vincristine, paclitaxel, docetaxel, foscarnet ,INH, etc..) in the last 6 months.
* Patients with evidence of metastasis at the initial assessment.
* Concomitant use of antioxidant vitamins (vitamin A, C, E),anticonvulsants, tricyclic antidepressants, other medications used for neuropathic pain (gabapentin, lamotrigine, carbamazepine).
* Presence of clinical evidence for severe cardiac illness (angina pectoris, uncontrolled hypertension, arrhythmias and left ventricular ejection fraction <50%).
* Preexisting peripheral neuropathy resulting from other causes such as diabetes and brain disorders, hypothyroidism, autoimmune diseases, hepatitis C.
* Patients with diabetes.
* Patients with inflammatory diseases (ulcerative colitis, rheumatoid arthritis).
* Patients with conditions associated with oxidative stress (smoking, tuberculosis, obesity).
* Patients with liver disease (fatty liver, hepatitis C, etc..).
* Patients who are candidates for monoclonal antibodies such as Trastuzumab and other targeted therapy (HER2 positive patients).
* Pregnant and breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-10-28 (Estimated); Primary Completion 2023-04-28 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
change in ejection fraction | 6 months
  Doxorubicin related cardiotoxicity will be assessed through :Echocardiography at baseline, Before starting the first chemotherapy cycle (baseline), after the last AC cycle (for assessment of N-terminal prohormone of brain naturetic peptide "NT-proBNP" ) and after the last doxorubicin/ cyclophosphamide (AC) cycle.
change in percentage of patients with peripheral sensory neuropathy | 6 months
  change in percentage of patients with peripheral sensory neuropathy grade ≥ 2 with the variation of both 12-item neurotoxicity questionnaire (Ntx-12) total score and pain rating scale score.

SECONDARY OUTCOMES:
changes in serum levels of the measured biological markers. | 6 months
  N-terminal prohormone of brain naturetic peptide "NT-proBNP" ) liver panel myeloperoxidase (MPO) neurofilament light chain (NFL) nuclear factor- Kabba B p65 (NF-ĸB p65) or TNF-alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Ibrahim AS, Khaled HM, Mikhail NN, Baraka H, Kamel H. Cancer incidence in egypt: results of the national population-based cancer registry program. J Cancer Epidemiol. 2014;2014:437971. doi: 10.1155/2014/437971. Epub 2014 Sep 21. PMID 25328522
- [Background] Klein I, Lehmann HC. Pathomechanisms of Paclitaxel-Induced Peripheral Neuropathy. Toxics. 2021 Sep 22;9(10):229. doi: 10.3390/toxics9100229. PMID 34678925
- [Background] Rawat PS, Jaiswal A, Khurana A, Bhatti JS, Navik U. Doxorubicin-induced cardiotoxicity: An update on the molecular mechanism and novel therapeutic strategies for effective management. Biomed Pharmacother. 2021 Jul;139:111708. doi: 10.1016/j.biopha.2021.111708. Epub 2021 May 13. PMID 34243633
- [Background] Huehnchen P, Muenzfeld H, Boehmerle W, Endres M. Blockade of IL-6 signaling prevents paclitaxel-induced neuropathy in C57Bl/6 mice. Cell Death Dis. 2020 Jan 22;11(1):45. doi: 10.1038/s41419-020-2239-0. PMID 31969555
- [Background] Cardinale D, Iacopo F, Cipolla CM. Cardiotoxicity of Anthracyclines. Front Cardiovasc Med. 2020 Mar 18;7:26. doi: 10.3389/fcvm.2020.00026. eCollection 2020. PMID 32258060
- [Background] Prasanna PL, Renu K, Valsala Gopalakrishnan A. New molecular and biochemical insights of doxorubicin-induced hepatotoxicity. Life Sci. 2020 Jun 1;250:117599. doi: 10.1016/j.lfs.2020.117599. Epub 2020 Mar 29. PMID 32234491
- [Background] Aboelwafa HR, El-Kott AF, Abd-Ella EM, Yousef HN. The Possible Neuroprotective Effect of Silymarin against Aluminum Chloride-Prompted Alzheimer's-Like Disease in Rats. Brain Sci. 2020 Sep 11;10(9):628. doi: 10.3390/brainsci10090628. PMID 32932753
- [Background] Abd Eldaim MA, Barakat ER, Alkafafy M, Elaziz SAA. Antioxidant and anti-apoptotic prophylactic effect of silymarin against lead-induced hepatorenal toxicity in rats. Environ Sci Pollut Res Int. 2021 Nov;28(41):57997-58006. doi: 10.1007/s11356-021-14722-8. Epub 2021 Jun 8. PMID 34100211
- [Background] Shokouhi G, Kosari-Nasab M, Salari AA. Silymarin sex-dependently improves cognitive functions and alters TNF-alpha, BDNF, and glutamate in the hippocampus of mice with mild traumatic brain injury. Life Sci. 2020 Sep 15;257:118049. doi: 10.1016/j.lfs.2020.118049. Epub 2020 Jul 4. PMID 32634430